CLINICAL TRIAL: NCT06826079
Title: Safety and Efficacy Study of Oral Sorbitol to Enhance the Therapeutic Effect of Neoadjuvant Chemotherapy Combined With Tirellizumab (PD-1 Inhibitor) in Patients With Locally Advanced Gastric Cancer
Brief Title: Safety and Efficacy Study of Sorbitol With Neoadjuvant Chemotherapy Combined With Tirellizumab (PD-1 Inhibitor) in Patients With Locally Advanced Gastric Cancer
Acronym: SNCCTGC
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Union01
Record Dates: First submitted 2025-02-09; First posted 2025-02-13 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Gastric Junction Adenocarcinoma; Gastric Cancer; Immunotherapy; Neoadjuvant Therapies
Keywords: sorbitol; tislelizumab; SOX; gastric cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Sorbitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- sorbitol (Experimental)
- placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Sorbitol — During the neoadjuvant treatment week, oral sorbitol 2-4g/ time, three times a day (with meals)
Other: Placebo — During the neoadjuvant treatment week, oral placebo 2-4g/ time, three times a day (with meals)
  Arms: placebo

SUMMARY:
The goal of this clinical trial is to learn if sorbitol works to enhance the therapeutic effect of neoadjuvant chemotherapy combined with Tirellizumab (PD-1 inhibitor) in patients with locally advanced gastric cancer. It will also learn about the safety of sorbitol. The main questions it aims to answer are:

Does sorbitol enhance the therapeutic effect of immunotherapy and increase the major response rate in patients with locally advanced gastric cancer? Does sorbitol with neoadjuvant chemotherapy combined with Tirellizumab (PD-1 inhibitor) can improve the prognosis of patients with locally advanced gastric cancer?

Researchers will compare sorbitol to a placebo (a look-alike substance that contains no drug) to see if sorbitol works to enhance the therapeutic effect of neoadjuvant chemotherapy combined with Tirellizumab (PD-1 inhibitor) in patients with locally advanced gastric cancer. .

Participants will:

Take sorbitol or a placebo every day for 3 months in 3 treatment cycles Visit the clinic once every 4 weeks for checkups and tests Keep a diary of their symptoms and the number of times they use a rescue inhaler Participants will follow up as planned until PD occurs, informed consent is withdrawn, or follow-up is lost (whichever occurs first). After the end of treatment and safety follow-up, all subjects will be followed up for survival (OS data collected every 3 months ±14 days)..

DETAILED DESCRIPTION:
1. Overall Design This study is an exploratory investigation on the efficacy of oral sorbitol combined with SOX chemotherapy and tislelizumab (PD-1 inhibitor) in the neoadjuvant treatment of advanced gastric/gastroesophageal junction adenocarcinoma based on the concepts of tumor metabolism and immunity. The study is divided into three phases: screening period, treatment period (neoadjuvant treatment, surgery and adjuvant treatment period), and follow-up period. A total of 100 subjects will be enrolled in this study and randomly divided into two groups. Group A: oral sorbitol + PD1 inhibitor + SOX for 3 cycles (1 cycle = every 3 weeks [Q3W]); Group B: placebo + PD1 inhibitor + SOX for 3 cycles (1 cycle = every 3 weeks [Q3W]) (see below for details).
2. Screening Period:

   Subjects must undergo screening and evaluation within 14 days before the first dose to determine their eligibility for the study. The specific criteria are: histologically confirmed, untreated HER2-negative gastric cancer or gastroesophageal junction (GEJ) cancer, with a clinical stage of cT3-4N+M0, and histological confirmation of mainly adenocarcinoma. Only Siewert type III and Siewert type II GEJ cancer patients who do not require combined thoracotomy are allowed to be enrolled. For patients who meet the inclusion and exclusion criteria, routine blood tests, imaging examinations, and Helicobacter pylori tests will be completed, and further molecular-level tests will be conducted, including MSI status, PD-1 expression CPS score, and EBER detection of pre-treatment biopsy pathological tissues.

   The enrolled subjects will be randomly divided into two groups. Group A: oral sorbitol + PD1 inhibitor + SOX for 3 cycles (1 cycle = every 3 weeks [Q3W]); Group B: oral placebo + PD1 inhibitor + SOX for 3 cycles (1 cycle = every 3 weeks [Q3W]).
3. Treatment Period

The treatment period will include the following phases:

1. Neoadjuvant treatment (before surgery) period: 3 cycles Group A (sorbitol diet group): PD1 inhibitor + SOX for 3 cycles (1 cycle = every 3 weeks [Q3W]); During the neoadjuvant treatment period, oral sorbitol 2-4g per dose, three times a day (with meals).

   Group B (placebo diet group): PD1 inhibitor + SOX for 3 cycles (1 cycle = every 3 weeks [Q3W]); During the neoadjuvant treatment period, oral placebo 2-4g per dose, three times a day (with meals).
2. Surgery: After evaluation of the efficacy of neoadjuvant treatment After neoadjuvant treatment, for subjects deemed eligible for surgery by the study, surgery should be performed within 2-6 weeks after the last dose of neoadjuvant treatment (including oral medication). For subjects who cannot undergo surgery, the subsequent treatment plan will be determined by the investigator based on the clinical situation. During the surgery, a small amount of pathological tissue should be taken and tested for AKR1B1/cGAS targets and sorbitol content.
3. Adjuvant treatment (after surgery) period: 5 cycles Adjuvant treatment stage: Unblinding after surgery, adjuvant treatment can start 3 weeks to 12 weeks after surgery (beyond 12 weeks, the investigator can decide whether to continue using the experimental drug). Subjects in Group A and Group B will be grouped according to TRG grading. Subjects with TRG scores of 0-1 will continue the original treatment plan, while those with TRG scores greater than 2 will only receive SOX chemotherapy for up to 5 cycles, or until the investigator determines that the subject has lost clinical benefit, died, is intolerant to toxicity, withdraws informed consent, or for other reasons specified in the protocol (whichever occurs first).

4. Follow-up Period: Including safety follow-up and survival follow-up. After the treatment ends, all subjects will be followed up. For subjects who discontinue treatment for reasons other than PD, follow-up will be conducted at the originally planned frequency until PD occurs, informed consent is withdrawn, or the subject is lost to follow-up (whichever occurs first). After the treatment ends and the safety follow-up is completed, all subjects will be followed up for survival (OS data will be collected every 3 months ± 14 days) until death, withdrawal of informed consent, loss to follow-up, or study termination (whichever occurs first).

ELIGIBILITY:
Inclusion Criteria

* Age: 18 years ≤ age ≤ 70 years, gender not restricted.
* Written informed consent obtained from the patient.
* Histologically confirmed, untreated HER2-negative gastric cancer or gastroesophageal junction (GEJ) cancer, with clinical stage cT3-4N+M0, and histological examination confirming mainly adenocarcinoma. Only Siewert type III GEJ cancer and Siewert type II GEJ cancer patients who do not require combined thoracotomy are eligible for inclusion.
* ECOG PS score of 0-1.
* Normal major organ function, meeting the following criteria:
* Blood routine examination criteria (no blood or blood product transfusion within 14 days, no use of G-CSF or other hematopoietic stimulating factors for correction):
* HB ≥ 90 g/L;
* ANC ≥ 1.5×109/L;
* PLT ≥ 125×109/L;
* Biochemical examination criteria:
* TBIL < 1.5ULN;
* ALT and AST < 2.5ULN, and for patients with liver metastasis, < 5ULN; serum Cr ≤ 1.25ULN or endogenous creatinine clearance rate > 50ml/min (Cockcroft-Gault formula);
* Fertile women must have taken reliable contraceptive measures or undergone a pregnancy test (serum or urine) within 7 days before enrollment, with a negative result, and be willing to use appropriate contraceptive methods during the trial and for 8 weeks after the last administration of the investigational drug. For men, they must agree to use appropriate contraceptive methods during the trial and for 8 weeks after the last administration of the investigational drug or have undergone surgical sterilization.

Exclusion Criteria

* Presence of distant organ metastasis and peritoneal disseminated metastasis.
* Active or previously recorded autoimmune or inflammatory diseases (including inflammatory bowel disease [such as colitis or Crohn's disease], diverticulitis [excluding diverticular disease], systemic lupus erythematosus, sarcoidosis syndrome, or Wegener's syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]), except for patients with vitiligo or alopecia, provided that they have celiac disease that can be controlled through diet after consultation with the study doctor.
* Other active malignant tumors within 5 years or concurrently. Patients with cured localized tumors, such as skin basal cell carcinoma, skin squamous cell carcinoma, superficial bladder cancer, prostate carcinoma in situ, cervical carcinoma in situ, breast carcinoma in situ, etc., can be included.
* Patients preparing for or having previously undergone organ or bone marrow transplantation.
* Uncontrolled concurrent diseases, including but not limited to: persistent or active infections (tuberculosis, HBV/HCV, pneumonia, etc.), symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, uncontrolled arrhythmia, active ILD, severe chronic gastrointestinal diseases with diarrhea, or conditions that may limit compliance with study requirements, significantly increase the risk of adverse events (AEs), or affect the ability of the subject to provide written informed consent.
* Patients currently using immunosuppressants, systemic or absorbable local hormones for immunosuppressive purposes (dose > 10mg/day prednisone or other equivalent efficacy hormones), and still using them within 2 weeks before enrollment.
* Patients who have previously received platinum-based, fluorouracil-based chemotherapy or targeted therapy, patients whose target lesions have undergone radiotherapy during combination therapy, or patients who have previously received other PD-1 antibody treatment or other PD-1/PD-L1 immune therapy.
* Have multiple factors that affect oral medication (such as inability to swallow, chronic diarrhea and intestinal obstruction, etc.);
* Have experienced significant clinically significant bleeding symptoms or have a clear bleeding tendency within the last three months, such as a history of black stool or hematemesis, or are at high risk of bleeding due to conditions such as intestinal perforation, gastric perforation, or extensive ulcers, or have active gastric ulcers and a positive fecal occult blood test (++) ;
* Have hypertension that cannot be well controlled with a single antihypertensive drug (systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg); have a history of unstable angina pectoris; have been newly diagnosed with angina pectoris within the last three months or have had a myocardial infarction within the last six months; have arrhythmia (including QTcF: male ≥ 450 ms, female ≥ 470 ms) and need long-term use of antiarrhythmic drugs or have New York Heart Association functional class ≥ II heart failure; Doppler ultrasound assessment: left ventricular ejection fraction (LVEF) < 50%;
* Urinalysis indicates proteinuria ≥ ++ and confirmed 24-hour urine protein quantification > 1.0 g;
* Have long-term non-healing wounds or incompletely healed fractures;
* Have abnormal coagulation function and a bleeding tendency (INR must be within the normal range without anticoagulants 14 days before enrollment); patients treated with anticoagulants or vitamin K antagonists such as warfarin, heparin or their analogues; low-dose warfarin (1 mg orally, once daily) or low-dose aspirin (daily dose not exceeding 100 mg) for prophylactic purposes is allowed if the international normalized ratio (INR) of prothrombin time is ≤ 1.5;
* Have experienced arterial or venous thrombotic events within the last year, such as cerebrovascular accidents (including transient ischemic attacks), deep vein thrombosis (except for venous thrombosis caused by previous chemotherapy catheterization and judged by the investigator to have healed), and pulmonary embolism, etc.;
* Have a history of abuse of psychotropic drugs and are unable to quit or have mental disorders;
* Have serious concomitant diseases that, in the judgment of the investigator, pose a significant risk to the patient's safety or affect the patient's ability to complete the study;
* Pregnant or lactating women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
major pathological response | From enrollment to the end of treatment at 3 months
pathological complete response | From enrollment to the end of treatment at 3 months

SECONDARY OUTCOMES:
objective response rate | From enrollment to the end of treatment at 3 months
R0 resection rate | From enrollment to the end of treatment at 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital Affiliated to Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No